CLINICAL TRIAL: NCT00702975
Title: A Phase II Study of Combination Therapy of Carboplatin -Gemcitabine Plus Bevacizumab Beyond Progression in Patients With Locally Advanced and/or Metastatic Non-small Cell Lung Cancer (NSCLC) Who Have Not Received Prior Systemic Therapy
Brief Title: Study of Combination Therapy of Carboplatin -Gemcitabine Plus Bevacizumab Beyond Progression in Patients With Locally Advanced and/or Metastatic Non-small Cell Lung Cancer (NSCLC) Who Have Not Received Prior Systemic Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULCN0107
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2012-04

CONDITIONS: Locally Advanced Non-Small Cell Lung Cancer; NSCLC
Keywords: phase II; NSCLC; bevacizumab; erlotinib; metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Carboplatin; Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Paclitaxel, Carboplatin and Bevacizumab,Erlotinib — 4 cycles (or less in case of progression) with carboplatin AUC 6 -paclitaxel 200mg/m2 -bevacizumab 15 mg/kg i.v. At (early) progress Bevacizumab 15 mg/kg i.v. q 21 days plus Erlotinib 150 mg/day orally
  Other Names: Carboplatin (L01XA02); Paxene (L01CD01); Avastin(L01XC07); Tarceva(L01XE03)

SUMMARY:
A phase II study of combination therapy of carboplatin -gemcitabine plus bevacizumab beyond progression in patients with locally advanced and/or metastatic non-small cell lung cancer (NSCLC) who have not received prior chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Advanced stage NSCLC (IIIB with malignant pleural effusion or stage IV excluding squamous cell histology, with measurable or evaluable disease.
* No prior systemic therapy for advanced NSCLC, prior therapy for early stage disease with one regimen is acceptable if it was completed at least 6 months prior to study entry.
* Palliative radiotherapy to painful bony metastases will be permitted prior to study entry if completed prior to initiation of study treatment, and there are no residual sequelae of therapy such as bone marrow suppression.
* Life expectancy of at least 3 months.
* ECOG Performance status 0-1 (see appendix 2)
* Age 18 or higher.
* Female patients with reproductive potential must have a negative serum pregnancy test within 72 hours prior to start of study medication. All female patients of childbearing potential, and all male patients, must agree to use a medically acceptable method of contraception or agree to be abstinent throughout the treatment period and for 3 months after discontinuation of treatment
* Patients must have normal organ and marrow function

Exclusion Criteria:

* Prior systemic treatment for advanced NSCLC. One prior regimen (up to 4 cycles) of neoadjuvant or adjuvant therapy for early stage disease will be allowed if completed at least 6 months prior to study entry.
* Known brain metastases (in case of clinical signs or symptoms of brain metastases radiological evaluation is mandatory).
* Prior treatment with bevacizumab or erlotinib.
* History of allergic reactions or sensitivity attributed to compounds of similar chemical or biologic composition to bevacizumab or erlotinib.
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in any other experimental drug study.
* Concomitant chemotherapy, radiotherapy or investigational agents.
* Evidence of bleeding diathesis or coagulopathy.
* Use of full dose anti-coagulant agents.
* Pregnant (positive pregnancy test) or lactating women.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to start, anticipation of need for major surgical procedure during the course of the study.
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to start.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to start.
* Serious, non-healing wound, ulcer, or bone fracture.
* Lung carcinoma of squamous cell histology or any histology in close proximity to a major vessel, or with significant cavitation as assessed by treating investigator in consultation with an attending radiologist.
* History of hemoptysis (bright red blood of 2.5 ml or more).
* Significant co-morbidities including:
* No uncontrolled hypertension (systolic > 150 mmHg and/or diastolic > 100 mmHg)
* Unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction within 6 months
* History of stroke within 6 months
* Clinically significant peripheral vascular disease
* Patients diagnosed with a trachea-oesophageal fistula
* Another active malignancy except for non-melanoma skin cancers in the last 5 years.
* Inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-09; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of erlotinib plus bevacizumab subsequent to the combination of carboplatin, paclitaxel and bevacizumab as determined by the maximum achieved disease control rate | at 18 weeks

SECONDARY OUTCOMES:
Efficacy of bevacizumab and erlotinib as determined by DCR; PFS; RR | at 6, 12 and 27 weeks

CONTACTS AND LOCATIONS:
Overall Officials: J. Timmer-Bonte, MD, Phd, Principal Investigator — UMCN st Radboud
Locations (1):
- University Lung Centre Nijmegen Dekkerswald, Groesbeek, Gelderland, Netherlands